CLINICAL TRIAL: NCT01684969
Title: Topical Haloperidol: Evidence of Absorption After Topical Administration
Brief Title: Evidence of Haloperidol Absorption After Topical Administration
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: lack of accrual and funding is about to expire.
Sponsor: Eric E. Prommer (Other)
Responsible Party: Sponsor-Investigator, Eric E. Prommer, Assistant Professor of Medicine, College of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-005661
Record Dates: First submitted 2012-03-19; First posted 2012-09-13 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Nausea; Vomiting
Keywords: Nausea; vomiting; gastrointestinal symptoms; palliative care
MeSH Terms: conditions — Nausea; Vomiting | interventions — Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- intravenous haloperidol (Active Comparator): intravenous haloperidol pharmacokinetics
  Interventions: Drug: Haloperidol
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Haloperidol — 0.5 mg iv x one dose
  Arms: intravenous haloperidol
Drug: Placebo — 0.5 mg iv , one dose
  Arms: Placebo

SUMMARY:
This will be a blinded study to compare the absorption of topical haloperidol with placebo

ELIGIBILITY:
Inclusion Criteria

* Age: patient must be 18 years or older and less than 70 years of age.
* Provision of informed consent
* No previous adverse reaction to haloperidol
* No current use of haloperidol
* Good health
* No alcohol within 24 hours of the study
* No significant cardiovascular, gastrointestinal, hematologic, neurologic, renal, hepatic or pulmonary disease.
* Normal neurologic exam

Exclusionary Criteria

* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the patient to participate in the study
* Recent cerebral trauma
* Study will exclude women who are pregnant and/or nursing
* Women who are of child bearing potential must have a negative urine pregnancy test.
* History of seizures
* Taking medications that can interact with haloperidol
* Subjects with significant cardiovascular (cardiac conduction deficits), gastrointestinal, hematologic, neurologic, renal, hepatic or pulmonary disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To measure the pharmacokinetics levels of haloperidol after topical administration compared with intravenous administration. | baseline to 240 minutes after administration.
  Measuring either the presence of absence of haloperidol

CONTACTS AND LOCATIONS:
Overall Officials: Eric Prommer, MD, Principal Investigator — Mayo Clinic